CLINICAL TRIAL: NCT03372694
Title: Clinical Study on the Effect of Comprehensive Rehabilitation Program Plus Chemotherapy Versus Chemotherapy on Quality of Life in Postoperative Non Small Cell Lung Cancer Patients With Stage IB-IIIA
Brief Title: Efficacy Study of Comprehensive Rehabilitation Program Plus Chemotherapy in Postoperative NSCLC Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Chest Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Shanghai Cancer Hospital, China (Other); Huadong Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHUTCM002
Record Dates: First submitted 2017-12-10; First posted 2017-12-14 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chemotherapy+Training+TCM (Experimental): Adjuvant Chemotherapy is performed within 6 weeks after operation. Rehabilitation training is mainly composed of gymnastic qigong, which will be started in one month after operation.
  Prescriptions formulated into granules origin from Professor Xu Ling in Yueyang hospital. Package of granules is made into four types with functions such as benefiting Qi recipe, benefiting Yin recipe, harmonizing stomach recipe, detoxication and resolving masses recipe. Patients will take harmonizing stomach recipe granules for the first week after chemotherapy and syndrome differentiation granules in TCM for second weeks from the end of chemotherapy. The patient will take TCM granules for 3 months.
  Interventions: Behavioral: Rehabilitation Training; Drug: TCM
- Chemotherapy+Education+TCM (Experimental): Adjuvant Chemotherapy is performed within 6 weeks after operation. Patients who received rehabilitation education will not accept rehabilitation training.
  Prescriptions formulated into granules origin from Professor Xu Ling in Yueyang hospital. Package of granules is made into four types with functions such as benefiting Qi recipe, benefiting Yin recipe, harmonizing stomach recipe, detoxication and resolving masses recipe. Patients will take harmonizing stomach recipe granules for the first week after chemotherapy and syndrome differentiation granules in TCM for second weeks from the end of chemotherapy. The patient will take TCM granules for 3 months.
  Interventions: Drug: TCM; Other: Rehabilitation Education
- Chemotherapy+Education+Placebo (Placebo Comparator): Adjuvant Chemotherapy is performed within 6 weeks after operation. Patients who received rehabilitation education will not accept rehabilitation training.
  Patients who received rehabilitation education will not accept rehabilitation training.
  We compromise the raw materials for the placebo including food color and artificial flavors. The placebo and therapeutic packages were stored in different cabinets, and only the dispensing technician knew the contents of the packages. The patient will take placebo granules for 3 months.
  Interventions: Other: Rehabilitation Education; Drug: placebo

INTERVENTIONS:
Behavioral: Rehabilitation Training — Patients will be trained in one month after operation. Rehabilitation training will be carried out between every two cycles of chemotherapy. Rehabilitation training is mainly composed of gymnastics qigong, which has long been regarded as a form of rehabilitation in Traditonal Chinese Medicine. According to the poor pulmonary function of patients with lung cancer after operation, Liu Zi Jue lung exercise is chosen to strengthen the pulmonary function of the human body in Chinese traditional health culture. Liu Zi Jue lung exercise intervention will be lead by an expert instructor, five times a week, 15 min/time.
  Other Names: gymnastics qigong; Liu Zi Jue lung exercises
  Arms: Chemotherapy+Training+TCM
Drug: TCM — four types with functions such as benefiting Qi recipe, benefiting Yin recipe, harmonizing stomach recipe and detoxication and resolving masses recipe. Each package contained 20g of water-soluble herbal granules that were manufactured at a Good Manufacture Practice standard facility (Tian Jiang Ltd, Jiangyin, China). Each package was labeled with a serial number. The prescription form comprised the stock list with both the name and serial number.
  Other Names: Prescriptions from Professor Xu Ling
  Arms: Chemotherapy+Education+TCM; Chemotherapy+Training+TCM
Other: Rehabilitation Education — General health education
  Other Names: health education
  Arms: Chemotherapy+Education+Placebo; Chemotherapy+Education+TCM
Drug: placebo — four types with functions such as benefiting Qi recipe, benefiting Yin recipe, harmonizing stomach recipe and detoxication and resolving masses recipe，with the same color, smell，taste, weight and package
  Other Names: control
  Arms: Chemotherapy+Education+Placebo

SUMMARY:
The investigators performed a multi-centered, randomized, placebo-controlled, prospective clinical trial on the effect of comprehensive rehabilitation program plus chemotherapy to improve quality of life(QOL) and long-term survival of postoperative non small cell lung cancer（NSCLC）patients with high risk stages IB to IIIA. The investigators plan to enroll 354 cases in 3 years (118 cases for chemotherapy plus rehabilitation training and traditional Chinese medicine (TCM), 118 cases for chemotherapy plus rehabilitation education and TCM,118 cases for chemotherapy plus rehabilitation education and placebo), expecting that comprehensive rehabilitation program plus chemotherapy has a better efficacy on improving QOL and long-term survival.

DETAILED DESCRIPTION:
NSCLC is one of the malignancies with high incidence and mortality. In recent years, surgery become the preferred treatment for early stage of NSCLC. Patients with high risk stages IB to IIIA may undergo radical surgery and complete 4-6 cycles of adjuvant chemotherapy. 5 year survival rate increased from 43.5% to 48.8%, but some patients will end chemotherapy because of the side effects of chemotherapy. Comprehensive rehabilitation program may alleviate the side effects as an effective treatment which including rehabilitation training and TCM.

The investigators performed a multi-centered, randomized, placebo-controlled, prospective clinical trial on the effect of comprehensive rehabilitation program plus chemotherapy to improve quality of life(QOL) and long-term survival of postoperative patients who need complete postoperative chemotherapy with high risk stages IB to IIIA. Patients are randomized into A observational group (chemotherapy plus rehabilitation training and TCM), B observational group(chemotherapy plus rehabilitation education and TCM) and control group (chemotherapy plus rehabilitation education and placebo). The treatment should be last three months and the patients will be followed up regularly. The primary efficacy assessments are: (1) QOL (QLQ-LC43 scale); (2) Pulmonary function test(PFTs): 1) Forced vital capacity (FVC); 2) Forced expiratory volume in one second (FEV1); 3) Forced expiratory flow rate from 25% to 50% (FEF25-50); 4) Residual volume (RV); 5) Total lung capacity (TLC). Secondary efficacy assessments are: (1) 2 years disease-free survival; (2) TCM symptoms changes; (3) Tumer markers (CEA, CA-125 and CYFRA21-1); (4) Exercise tolerance; (5) Toxicity, side effects and security of the treatments will be assessed at the same time. The investigators plan to enroll 354 cases in 3 years (118 cases for chemotherapy plus rehabilitation training and traditional Chinese medicine (TCM), 118 cases for chemotherapy plus rehabilitation education and TCM,118 cases for chemotherapy plus rehabilitation education and placebo), expecting that comprehensive rehabilitation program plus chemotherapy has a better efficacy on improving QOL and long-term survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with completely resected stage IB-IIIA non-small-cell lung cancer who will receive chemotherapy for the first time within 6 weeks after the operation.
* Between the ages of 18 to 75 years old;
* The score of ECOG ≥2 points
* Without major organ dysfunction: hemoglobin ≥10 g/dL, absolute neutrophil count (ANC) ≥1.5*10^9/L, platelets ≥100 *10^9/L; normal hepatic and renal function

Exclusion Criteria:

* Indefinite pathological diagnosis;
* Expected survival time < 6 months
* Combined with heart, liver, kidney and hematopoietic system and other serious diseases
* The patient was treated with antibiotics or infected one week before the test;
* Pregnant or child breast feeding women;
* Mental or cognitive disorders;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Quality of life (QOL) | Time Frame: baseline, at 4 months
  QOL is assessed using European Organization for Research and Treatment of Cancer Quality of Life QuestionnaireLung Cancer 43 (EORTC QLQ-LC43).

SECONDARY OUTCOMES:
Residual capacity (RV) | after intervention at 2 weeks
  RV is measured in a test known as Lung valume(LV)spirometry,a type of pulmonary function test.RV is the volume of air remaining in the lungs after a maximal expiratory effort.
Total lung capacity（TLC） | after intervention at 2 weeks
  TLC is measured in a test known as Lung valume(LV)spirometry,a type of pulmonary function test.TLC equals the vital capacity plus the residual capacity.
Forced vital capacity (FVC) | after intervention at 2 weeks
  FVC is the volume of air exhaled with maximum effort and speed after a full inspiration. FVC is measured in a test known as spirometry, a type of pulmonary function test.
Forced expiratory volume in one second(FEV1) | after intervention at 2 weeks
  FEV1 is an individual test measure used to assess limitations in airflow, a type of pulmonary function test,which measures the amount of air exhaled in onesecond.
Maximum mid expiratory flow(MMEF) | after intervention at 2 weeks
  MMEF is forced expiratory flow between 25% and 75% of forced vital capacity,a type of pulmonary function test.
Disease-free survival (DFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Time from randomization to first recurrence or metastasis
TCM symptoms changes | after intervention at 4 months
  TCM symptoms changes are according to the lung cancer symptom classification quantization table in "Guiding Principles for Clinical Research of Traditional Chinese Medicine in the Treatment of Lung Cancer (2002 Edition)"
Tumor markers | after intervention at 4 months
  Tumor markers include CEA, CA-125 and CYFRA21-1
Safety assessment evaluated according to Common Toxicity Criteria | after intervention at 4 months
  Safety assessment is evaluated according to Common Toxicity Criteria (CTC 3.0)

CONTACTS AND LOCATIONS:
Overall Officials: Ling Xu, MD & PhD, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- YueYang Hosptial of Intergrated Traditional Chinese and Western Medicine,Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang YL, Jiao LJ, Gong YB, Xu JF, Ni J, Shen XY, Zhang J, Zhou D, Qian CX, Wang Q, Yao JL, Yang WX, Su LZ, Wang LY, Li JQ, Yao YQ, Zhang YH, Wang YC, Chen ZW, Xu L. Patient-Reported Outcomes of Postoperative NSCLC Patients with or without Staged Chinese Herb Medicine Therapy during Adjuvant Chemotherapy (NALLC 2): A Randomized, Double-Blind, Placebo-Controlled Trial. Chin J Integr Med. 2024 Nov;30(11):963-973. doi: 10.1007/s11655-024-4114-9. Epub 2024 Sep 12. PMID 39266862
- [Derived] Yao J, Jiao L, Yao Y, Lu Y, Shi J, Li J, Chen P, Xu L, Gong Y. The effect of comprehensive rehabilitation program plus chemotherapy on quality of life in patients with postoperative non-small-cell lung cancer: study protocol of a multicenter randomized clinical trial. Trials. 2020 Apr 3;21(1):309. doi: 10.1186/s13063-020-4162-1. PMID 32245480